CLINICAL TRIAL: NCT07365046
Title: Comprehensive Analysis of the Swallowing Mechanism Using High-resolution Manometry With Impedance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-Manometry
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Extraesophageal Reflux; Laryngopharyngeal Reflux; Dysphagia; Chronic Cough
Keywords: Extraesophageal reflux; Laryngopharyngeal reflux; Dysphagia; Chronic cough; high-resolution manometry; 24-hour pH-impedance monitoring
MeSH Terms: conditions — Laryngopharyngeal Reflux; Deglutition Disorders; Chronic Cough | interventions — Electric Impedance

STUDY DESIGN:
Masking Description: No masking will be used in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extraoesophageal reflux (Experimental): Patients with extraoesophageal reflux will be enrolled in this study arm.
  Interventions: Diagnostic Test: High resolution oesophageal manometry with impedance; Diagnostic Test: 24-hour pH metry
- Dysphagia (Experimental): Patients with dysphagia reflux will be enrolled in this study arm.
  Interventions: Diagnostic Test: High resolution oesophageal manometry with impedance

INTERVENTIONS:
Diagnostic Test: High resolution oesophageal manometry with impedance — Patients with extraoesophageal reflux and dysphagia will undergo high resolution oesophageal manometry with impedance.
Diagnostic Test: 24-hour pH metry — Patients with extraoesophageal reflux will undergo 24-hour pH-metry.
  Arms: Extraoesophageal reflux

SUMMARY:
The aim of this project is to perform a detailed evaluation of upper esophageal sphincter function and the swallowing mechanism in patients with swallowing disorders or suspected extraesophageal reflux using high-resolution manometry with impedance and 24-hour pH-impedance monitoring.

DETAILED DESCRIPTION:
The project seeks to improve diagnostic accuracy, identify functional abnormalities that are not detectable by conventional diagnostic methods, and establish a foundation for more effective and targeted therapeutic strategies.

The upper esophageal sphincter (UES) represents a crucial functional structure at the junction of the digestive and respiratory tracts. Its proper function is essential for the coordination of the swallowing process and for the protection of the upper airways. Disorders of the UES may be associated with a wide range of otorhinolaryngological symptoms, including dysphagia, globus pharyngeus, chronic cough, hoarseness, laryngeal dysfunction, and voice disorders. Modern diagnostic techniques, such as 24-hour esophageal impedance monitoring and high-resolution manometry (HRM), enable detailed assessment of gastroesophageal reflux and esophageal pressure dynamics, thereby offering new possibilities for the diagnosis and understanding of these conditions.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* patients with swallowing difficulties suspected of having a functional oesophageal disorder or patients with clinical signs of extra-oesophageal reflux (Reflux Symptom Index [RSI] ≥ 13 or Reflux Symptom Score-12 [RSS-12] ≥ 11) signed informed consent

Exclusion Criteria:

* patients with a diagnosed tumor of the esophagus or upper airway, or with strong clinical suspicion of a tumor of the esophagus or upper airway
* severe neurological disease affecting swallowing
* pregnancy
* surgery involving the head, neck, or esophagus within the last 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
PAET (Proximal Acid Exposure Time) | 24 hours
  PAET (Proximal Acid Exposure Time) - acid exposure to the proximal oesophageus will be measured in per cent of the whole 24-h period.
Upper esophageal sphincter (UES) Integrated Relaxation Pressure (IRP) | 15 minutes
  UES IRP is a measure of the extent of UES relaxation measured in mmHg
UES Maximum Admittance | 15 minutes
  UES MaxAd is the highest admittance value recorded during trans-sphincteric bolus flow measured in milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Tichý, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon reasonable request.

REFERENCES:
- [Background] Omari TI, Maclean JCF, Cock C, McCulloch TM, Nativ-Zeltzer N, O'Rourke AK, Szczesniak MM, Wu PI, Allen J, Aoyagi Y, Bayona HHG, Carrion S, Ciucci MR, Davidson K, Dhar SI, Hamdy S, Howell R, Jones C, Knigge MA, Moonen A, Postma GN, Puntil-Sheltman J, Rameau A, Regan J, Schar M, Rommel N. Defining Pharyngeal and Upper Esophageal Sphincter Disorders on High-Resolution Manometry-Impedance: The Leuven Consensus. Neurogastroenterol Motil. 2025 Apr 9:e70042. doi: 10.1111/nmo.70042. Online ahead of print. PMID 40202098
- [Background] Omari T, Cock C, Wu P, Szczesniak MM, Schar M, Tack J, Rommel N. Using high resolution manometry impedance to diagnose upper esophageal sphincter and pharyngeal motor disorders. Neurogastroenterol Motil. 2023 Jan;35(1):e14461. doi: 10.1111/nmo.14461. Epub 2022 Sep 19. PMID 36121685
- [Background] Wang YC, Wang CC, Chuang CY, Tsou YA, Peng YC, Chang CS, Lien HC. Baseline Impedance via Manometry Predicts Pathological Mean Nocturnal Baseline Impedance in Isolated Laryngopharyngeal Reflux Symptoms. J Neurogastroenterol Motil. 2025 Jan 31;31(1):63-74. doi: 10.5056/jnm24051. PMID 39779205
- [Background] Watson W, Simmons E, Adebowale A, Banda C, Qu R, Becerra B, Crawley B, Murry T, Krishna P. Manometric Abnormalities in Patients With and Without Chronic Cough. Am J Otolaryngol. 2024 Nov-Dec;45(6):104445. doi: 10.1016/j.amjoto.2024.104445. Epub 2024 Jul 31. PMID 39102762
- [Background] Tseng WH, Hsu WC, Hsiao TY, Wu JF, Lee HC, Wang HP, Wu MS, Tseng PH. Anatomical and physiological characteristics in patients with Laryngopharyngeal Reflux Symptoms: A case-control study utilizing high-resolution impedance manometry. J Formos Med Assoc. 2022 Jun;121(6):1034-1043. doi: 10.1016/j.jfma.2021.07.025. Epub 2021 Aug 6. PMID 34366184